CLINICAL TRIAL: NCT01520532
Title: Evaluate Reduction in Asymptomatic Cerebral Embolism
Brief Title: Evaluation of the Incidence of Cerebral Lesions Post Pulmonary Vein Ablation Catheter (PVAC)
Acronym: ERACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MDT-AFS-ERACE
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ablation (Other)
  Interventions: Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — MRI's will be performed on all subjects at Enrollment and Pre-Discharge (Post Ablation). Subjects with a positive MRI (cerebral lesion) at the Pre-Discharge will undergo an MRI at the 1 month follow-up visit.

SUMMARY:
The purpose of the study is to determine the rate of diffusion weighted (DW)-MRI cerebral lesions following a Pulmonary Vein Ablation Catheter (PVAC) ablation procedure performed using best practices, including optimized procedural techniques and anti-coagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old
* Subject has been diagnosed with atrial fibrillation (AF)
* Subject is indicated for a pulmonary vein ablation using PVAC
* Subject (or subject's legally authorized representative) is able and and willing to give informed consent.

Exclusion Criteria:

* Subject has permanent AF
* Subject has a left atrial thrombus detected on TEE
* Subject has had a prior left atrial ablation
* Subject has a intracardiac thrombus
* Subject is contraindicated for Warfarin (Coumadin)
* Subject has a cardiac valve prosthesis
* Subject has a significant congenital heart defect corrected or not including atrial septal defects or pulmonary vein abnormalities but not including minor PFO)
* Subject has presence of any pulmonary vein stents
* Subject has presence of any pre-existing pulmonary vein stenosis
* Subject has had a cerebral ischemic event (strokes or transient ischemic attacks [TIA]) which occurred during the 6 month interval preceding the Consent Date
* Subject is a woman known to be pregnant
* Subject is unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves De Greef, MD, Principal Investigator — AZ Middelheim; Lucas Boersma, MD, Principal Investigator — AZ Sint Antonius Ziekenhuis; Thomas Deneke, MD, Principal Investigator — Krankenhaus Porz am Rheim; Stefano Nardi, MD, Principal Investigator — Pineta Grande Hospital; Atul Verma, MD, Principal Investigator — Southlake Regional health Center; Stefan G Spitzer, MD, Principal Investigator — Praxisklinik Herz- und Gefässe; Philippe Debruyne, MD, Principal Investigator — Imelda Hospital, Bonheiden
Locations (7):
- Belgium (2):
  - AZ Middelheim, Antwerp
  - Imelda Ziekenhuis, Bonheiden
- Southlake Regional Health Center, Newmarket, Ontario, Canada
- Germany (2):
  - Herz- und Gefäß-Klinik, Bad Neustadt/Saale
  - Praxisklinik - Herz- und Gefässe, Dresden
- Clinica Pineta Grande, Castel Volturno, Italy
- AZ Sint Antonius Ziekenhuis, Nieuwegein, Netherlands

REFERENCES:
- [Result] Verma A, Debruyne P, Nardi S, Deneke T, DeGreef Y, Spitzer S, Balzer JO, Boersma L; ERACE Investigators. Evaluation and reduction of asymptomatic cerebral embolism in ablation of atrial fibrillation, but high prevalence of chronic silent infarction: results of the evaluation of reduction of asymptomatic cerebral embolism trial. Circ Arrhythm Electrophysiol. 2013 Oct;6(5):835-42. doi: 10.1161/CIRCEP.113.000612. Epub 2013 Aug 27. PMID 23983245

RESULTS

PARTICIPANT FLOW:
Groups:
- Ablation: Single-arm study, all subjects received a radio-frequency (RF) ablation with the goal of achieving Pulmonary Vein Isolation (PVI).
Period: Overall Study
Arm/Group | Ablation
Started | 60 (Subjects who underwent an ablation and had post-procedure MRI)
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ablation
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 41
Region of Enrollment [Number; unit: participants]
  Canada | 12
  Belgium | 13
  Germany | 12
  Netherlands | 12
  Italy | 11

OUTCOME MEASURES:

1. Primary Outcome: New Asymptomatic Cerebral Embolic Lesions, Visualized as 'Bright Spots' on Post-ablation MRI.
Description: An acute embolic lesion is defined as a focal hyper-intense area detected on the diffusion-weighted (DW) sequence, corresponding to a hyper-intense signal intensity in the fluid-attenuated inversion recovery (FLAIR) sequence, and also confirmed by apparent diffusion coefficient (ADC) mapping to rule out a shine-through artifact.
Time Frame: Within 1-3 days post ablation
Population: All subject who underwent an ablation and post-procedure MRI.
Measure: Number; unit: participants
Arm/Group | Ablation
Number analyzed (Participants) | 60
participants | 1

2. Secondary Outcome: Acute Safety Events
Description: Assess the number of procedure or device-related serious adverse events when applying best practices with PVAC.
Time Frame: 30 days
Population: All subjects who underwent an ablation and post-procedure MRI
Measure: Number; unit: events
Arm/Group | Ablation
Number analyzed (Participants) | 60
events | 1

3. Secondary Outcome: Acute Efficacy, as Determined by Complete Pulmonary Vein Isolation (PVI) Per Subject.
Description: The number of subjects with pulmonary vein isolation (PVI) at the end of ablation procedure. This will characterize if use of best practices during PVAC ablation negatively affects acute efficacy.
Time Frame: Day 1 (End of Procedure)
Population: All subjects who underwent ablation and post-procedure MRI.
Measure: Number; unit: participants
Arm/Group | Ablation
Number analyzed (Participants) | 60
participants | 60

ADVERSE EVENTS:
Arm/Group | Ablation
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 11/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation (N=60)
Bleeding (Vascular disorders) | 1 (1) — Groin bleed requiring intervention (thrombin administration)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation (N=60)
Groin Bleed (Vascular disorders) | 11 (11) — Mild groin bleed at location of sheath insertion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less